CLINICAL TRIAL: NCT02205658
Title: Standardization of the Adult/ Adolescent Sensory History
Brief Title: Sensory Processing Difficulties in Adults and Adolescents
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Spiral Foundation at OTA Watertown (Other)
Collaborators: Maxwell Hurston Charitable Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1027
Record Dates: First submitted 2014-07-29; First posted 2014-07-31 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Sensory Processing Dysfunction
Keywords: Sensory Processing; Autism
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Autism: Individuals, aged 18-95 years, with a pre-existing diagnosis of Autism Spectrum Disorder with or without a co-morbid diagnosis of Sensory Processing Disorder.
- Sensory Processing: Individuals, aged 18-95 years, with a pre-existing diagnosis of Sensory Processing Disorder with no co-morbid diagnosis of Autism Spectrum Disorder
- Typical: Typically functioning individuals aged 13-95 years

SUMMARY:
The purpose of this study is to establish normative data for the Adult/Adolescent Sensory History (ASH) and to determine if the ASH is able to discriminate between individuals aged 13-95 years, with Autism Spectrum Disorder (ASD) with or without co-morbid Sensory processing Disorder (SPD), individuals with SPD with no co-morbid ASD, and individuals who are typically functioning.

It is anticipated that individuals with ASD will have the most problems with sensory processing, those with SPD will also have problems in comparison to typical individuals. It is also hypothesized that the measure will be able to discriminate between the three groups.

ELIGIBILITY:
Inclusion Criteria:

* Autism and Sensory Processing groups aged 18-95 years, Typical group aged 13-95 years
* Have no self-reported diagnosed neurological motor coordination problem (e.g. cerebral palsy)
* Have no mental health diagnoses involving psychosis (e.g. manic-depression or schizophrenia)
* Be able to read and speak sufficient English as survey is only available in English.

Exclusion Criteria:

* Outside of the designated age range
* Unable to complete the survey independently

Ages: 13 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals will be a nationally representative sample of US residents
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-09 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Sensory processing difficulties | 15-20 minutes
  This study proposes to measure sensory processing problems by self report

CONTACTS AND LOCATIONS:
Overall Officials: Teresa A May Benson, ScD, Principal Investigator — The Spiral Foundation
Locations (1):
- The Spiral Foundation, Newton, Massachusetts, United States

REFERENCES:
- See also: Spiral Foundation website — http://www.thespiralfoundation.org